CLINICAL TRIAL: NCT00738023
Title: Free Fatty Acid-Induced Hypertension in Obese Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Guillermo Umpierrez, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 967-2003
Record Dates: First submitted 2008-08-19; First posted 2008-08-20 (Estimated); Results first posted 2014-12-30 (Estimated); Last update posted 2014-12-30 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes; Hypertension
Keywords: diabetes,; hypertension,; free-fatty acids
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Hypertension; Diabetes Mellitus | interventions — Rosiglitazone; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Diabetics (Active Comparator): Obese, normotensive African-Americans with diabetes received Intralipid 20% at 40ml/hr intravenously for 48 hours, then normal saline 0.9% at 40 ml/hr intravenously for 48 hours, and then randomized to rosiglitazone for six weeks followed by Intralipid 20% at 40ml/hr intravenously for 48 hours
  Interventions: Drug: Rosiglitazone; Drug: Normal saline 0.9%; Drug: Intralipid 20%
- Non-Diabetic (Active Comparator): Obese, normotensive African-Americans without diabetes received Intralipid 20% at 40ml/hr intravenously for 48 hours
  Interventions: Drug: Intralipid 20%

INTERVENTIONS:
Drug: Rosiglitazone — Diabetic subjects will be receive rosiglitazone for 6 weeks
  Arms: Diabetics
Drug: Normal saline 0.9% — Normal saline 0.9% intravenous infusion at 40ml/hr for 48 hours
  Arms: Diabetics
Drug: Intralipid 20% — Intralipid 20% at 40ml/hr intravenously for 48 hours

SUMMARY:
Insulin resistance has been implicated as the central pathogenetic feature of cardiovascular risk factor cluster that includes hypertension, impaired glucose tolerance, diabetes, dyslipidemia, and hemostatic disorders. Recent evidence suggests that increased levels of free fatty acids (FFA) in obese subjects is a leading candidate in the pathogenesis of insulin resistance (1-4). In our preliminary studies on the effect of FFA on insulin secretion and action (lipotoxicity), we have observed that the infusion of Intralipid/heparin to increase FFA ~ four-fold-baseline levels for 48 hours results in a significant and reproducible raise in systolic and diastolic blood pressure (BP) in obese African American subjects with and without diabetes. The increase in blood pressure is apparent after 12 hours of infusion, reaching a peak increment of 32 mm Hg in systolic and 14 mm Hg in diastolic pressure at 24 hours. These preliminary findings indicate that, in addition to the well-known effect on insulin resistance, sustained elevation of FFA results in the development of an acute metabolic syndrome.

DETAILED DESCRIPTION:
The FFA-induced hypertension constitutes a useful model with which to examine disease mechanisms and test new therapeutic interventions to correct the different disorders associated with insulin resistance and metabolic syndrome. The effect of FFA on insulin action is well established (4-6); however, the pressor effect of FFA infusion in obese subjects has not been investigated. We hypothesize that observed changes in blood pressure is the result of acute endothelial dysfunction due to increased FFA concentration; and that rosiglitazone, a PPAR gamma receptor agonist, will protect against FFA-induced elevation in blood pressure and endothelial dysfunction in obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 18 and 70 years.
* Subjects must have a BMI of ≥ 30 kg/m2.
* Subjects must have a BP < 130/80 mm Hg and no prior history of hypertension.
* A known history of type 2 diabetes mellitus < 3 years (now 5 years).
* Subjects must have an HbA1c of < 9%.
* Diabetic subjects must have been receiving as their only current anti-diabetic therapy stable doses of sulfonylureas for the last 2 months.
* Subjects must be able to understand and willing to adhere to the study protocol.

Exclusion Criteria:

* Subjects with history of hypertension (BP > 140/90 mm HG) or who have received antihypertensive drug therapy prior to the study.
* Obese nondiabetic controls with impaired glucose tolerance (2-hour glucose between 140 - 199 mg/dl) during a 75-g OGTT.
* Diabetic subjects who require insulin therapy or have received an insulin sensitizer agent (metformin, rosiglitazone, pioglitazone) within 3 months of entering the study (at SV1, week-2).
* Subjects with fasting triglyceride levels > 250 mg/dL prior to the study (at SV1, week-2).
* Clinically relevant hepatic disease (ALT 2.5x > upper limit of normal), or other significant medical or surgical illness.
* Renal failure, as shown by a serum creatinine ≥1.5 mg/dL for males, or ≥ 1.4 mg/dL for females.
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study.
* Female subjects are pregnant or breast feeding at time of enrollment into the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-03; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (1):
- Grady Memorial Hospital, Atlanta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Four subjects were withdrawn due to exclusion criteria prior to randomization. Non-diabetic arm did not continue after the first intralipid infusion (period 1).
Groups:
- Diabetics: Obese, normotensive African-Americans with diabetes received Intralipid 20% at 40ml/hr intravenously for 48 hours, normal saline 0.9% at 40 ml/hr intravenously for 48 hours, and rosiglitazone for six weeks followed by Intralipid 20% at 40ml/hr intravenously for 48 hours
Period: Intralipid Infusion
Arm/Group | Diabetics | Non-Diabetic
Started | 19 | 13
Completed | 19 | 13
Not Completed | 0 | 0
Period: Saline Infusion
Arm/Group | Diabetics | Non-Diabetic
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0
Period: Intralipid Infusion (Post 6 Wks of Drug)
Arm/Group | Diabetics | Non-Diabetic
Started | 19 | 0
Completed | 19 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Diabetics: Obese, normotensive African-Americans with diabetes received Intralipid 20% at 40ml/hr intravenously for 48 hours, normal saline 0.9% at 40 ml/hr intravenously for 48 hours, and rosiglitazone for 6 weeks followed by Intralipid 20% at 40ml/hr intravenously for 48 hours
- Non-Diabetic: Obese, normotensive African-Americans without diabetes received Intralipid 20% at 40ml/hr intravenously for 48 hours and normal saline 0.9% at 40 ml/hr intravenously for 48 hours
- Total: Total of all reporting groups
Arm/Group | Diabetics | Non-Diabetic | Total
Number analyzed (Participants) | 19 | 13 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 41 (2) | 42 (1) | 41.5 (0.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 16
  Male | 12 | 4 | 16

OUTCOME MEASURES:

1. Primary Outcome: Changes in Systolic Blood Pressure During Initial Intralipid Infusion
Description: Systolic blood pressure change from baseline during an 48-hour intralipid infusion
Time Frame: Baseline, 48 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Diabetics | Non-Diabetic
Number analyzed (Participants) | 19 | 13
mmHg | 23 (9) | 13 (12)

2. Secondary Outcome: Changes in Systolic Blood Pressure During Saline Infusions
Description: Systolic blood pressure change from baseline during an 48-hour normal saline infusion in obese diabetic subjects
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Diabetics
Number analyzed (Participants) | 19
mmHg | 0 (4)

3. Secondary Outcome: Changes in Systolic Blood Pressure During Intralipid Infusion Post-rosiglitazone Intervention
Description: Systolic blood pressure change from baseline during an 48-hour intralipid infusion after taking rosiglitazone for 6 weeks in obese diabetic subjects
Time Frame: 48 hours
Measure: Mean (Standard Error); unit: mmHg
Arm/Group | Diabetics
Number analyzed (Participants) | 19
mmHg | 1 (6)

ADVERSE EVENTS:
Arm/Group | Diabetics | Non-Diabetic
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/13
Other Adverse Events (participants affected / at risk) | 2/19 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Diabetics (N=19) | Non-Diabetic (N=13)
pain at IV site (Vascular disorders) | 2 (2) | 1 (1) — mild irritation of the vein at the infusion site for intralipid

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No